CLINICAL TRIAL: NCT02506855
Title: Intraoperative Transversus Abdominis Plane Block for Gynecologic Surgery (GYNTAP): Modifying an Existing Technique for Ease of Administration and Increased Accuracy
Brief Title: Intraoperative Transversus Abdominis Plane Block for Gynecologic Surgery (GYNTAP)
Acronym: GYNTAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The investigator decided not to continue the study.
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Mildred Ridgway, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014-0238
Record Dates: First submitted 2015-06-11; First posted 2015-07-23 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Study participants will undergo intraoperative transversus abdominis plane (TAP) block with the syringe of medication supplied by the pharmacy using a syringe with attached spinal needle between the transversus abdominis and internal oblique. The spinal needle will be threaded horizontally and as far laterally at the superior aspect of the vertical axis of the incision as possible within this space and anesthetic will be injected after an initial pull back on the syringe to ensure there is no arterial exposure as per the following schedule:
  Weight <70kg: Ropivacaine 75mg - 150 mg on each side (20mL ropivacaine 3.75mg/ml each side)
  Weight greater than or equal to 70kg: Ropivacaine 100mg - 200mg on each side (20mL ropivacaine 5mg/ml each side
  Interventions: Drug: Ropivacaine; Procedure: Transversus Abdominis Plane Block
- Group B (Placebo Comparator): Study participants will undergo intraoperative transversus abdominis plane (TAP) block with the syringe of medication supplied by the pharmacy using a syringe with attached spinal needle between the transversus abdominis and internal oblique. The spinal needle will be threaded horizontally and as far laterally at the superior aspect of the vertical axis of the incision as possible within this space and the placebo solution will be injected after an initial pull back on the syringe to ensure there is no arterial exposure as per the following schedule:
  Weight <70kg: 20mL each side
  Weight greater than or equal to 70kg: 20mL each side
  Interventions: Other: Placebo; Procedure: Transversus Abdominis Plane Block

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Group A
Other: Placebo
  Arms: Group B
Procedure: Transversus Abdominis Plane Block

SUMMARY:
This study attempts to learn about the effectiveness of a modification to the Transversus Abdominis Plane (TAP) block that works by anaesthetizing the sensory afferents of the abdominal wall postoperatively using ultrasound guidance. The investigators want to see if regional blocks placed by the surgeon intraoperatively to assure regional anesthetic spread in the appropriate plane could reduce error and improve postoperative recovery.

DETAILED DESCRIPTION:
This study is a prospective, randomized blinded study that investigates the efficacy of a transversus abdominis plane block under direct view. In this pilot study involving gynecologic patients undergoing open (abdominal wall incision either vertically or horizontally) hysterectomy or other related gynecologic surgery, the investigators will use ropivacaine versus saline for the placebo control group, which in both groups involves injection of agent directly into the appropriate fascial layers prior to abdominal wall closure. Efficacy is to be assessed via measurement of pain scores, nausea and vomiting, and opioid consumption in both participant groups. The number of dermatomes which are blocked in both participant groups during the first 24 hours following surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old and not pregnant
* Must be able to provide informed consent - functional understanding of English
* Undergoes exploratory laparotomy with midline abdominal incision

Exclusion Criteria:

* History of substance abuse
* History of chronic pain syndrome
* Daily opioid use for more than 1 month
* Patients considered to have chorioamnionitis at the time of cesarean surgery as determined by the attending physician
* Prior abdominal surgery involving mesh or placement of an ostomy site as this may disrupt the plane in which the anesthetic may spread
* Allergy to local anesthetics
* History of cardiac arrhythmias or cardiac abnormalities
* History of seizure disorder
* Liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Milligrams of Diludid Consumption During First 48 hours Following Surgery | 48 hours postoperatively
  The amount of diludid received per participant will be recorded from participant medication record at the specified time frame.

SECONDARY OUTCOMES:
Level of Nerve (Dermatome) Block | 4hrs postoperative and on postoperative day 1
  The investigator will complete dermatomal assessments at the specified time frames by using a stimulus in the area of the transversus abdominis plane block to determine the effectiveness of the block.
Pain Scores at Rest and with Movement | 2, 4, 6, 12, 24, 36 and 48 hours postoperatively.
  Pain severity will be measured using a validated Numerical Rating Scale with 0cm=no pain and 10cm=worst pain imaginable.
Postoperative Nausea and Vomiting | 2, 4, 6, 12, 24, 36 and 48 hours postoperatively.
  Nausea will be measured using a validated postoperative nausea and vomiting scale known as the Impact Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States